CLINICAL TRIAL: NCT06959186
Title: High-Frequency QRS and Fibrosis Biomarkers for Risk Stratification in Chronic Heart Failure: A Multicenter Prospective Cohort Study
Brief Title: Risk Stratification Via HF-QRS and Fibrosis Biomarkers in Heart Failure
Acronym: STRIVE
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: BBMUFH20250428
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Myocardial Fibrosis; high-frequency QRS; biomarker; rehospitalization; mortality
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Heart Failure Patients: Participants diagnosed with chronic heart failure (CHF), classified based on left ventricular ejection fraction (LVEF) into heart failure with reduced ejection fraction (HFrEF), heart failure with mildly reduced ejection fraction (HFmrEF), or heart failure with preserved ejection fraction (HFpEF) groups. All participants receive standard-of-care heart failure management according to clinical guidelines. No investigational intervention is assigned; this is an observational cohort.

SUMMARY:
This study aims to evaluate whether high-frequency QRS (HF-QRS) signal parameters and circulating myocardial fibrosis biomarkers (such as PIIINP, Galectin-3, and sST2) can improve risk stratification in patients with chronic heart failure (CHF). In this prospective, multicenter cohort study (STRIVE cohort), patients with CHF will be enrolled and followed for 18 months. Clinical data, routine heart function measures (such as NT-proBNP and LVEF), HF-QRS features from standard 12-lead ECG, and serum fibrosis biomarker levels will be collected. The study will assess the association of HF-QRS abnormalities and fibrosis biomarker levels with major clinical outcomes, including cardiovascular mortality, first heart failure-related rehospitalization, malignant arrhythmia events, all-cause rehospitalization and mortality. By integrating electrophysiological and molecular markers, this research aims to develop a novel, non-invasive predictive model to support early risk identification and personalized management of heart failure patients.

DETAILED DESCRIPTION:
Heart failure (HF) remains a leading cause of morbidity, hospitalization, and mortality worldwide. Traditional risk assessment tools, such as left ventricular ejection fraction (LVEF) and NT-proBNP levels, are widely used but have limitations in early identification of high-risk patients, particularly those with subclinical myocardial injury or conduction abnormalities. Recent advances suggest that high-frequency QRS (HF-QRS) signal abnormalities extracted from standard 12-lead ECGs can sensitively detect microstructural myocardial changes, such as fibrosis and conduction disruption, earlier than conventional markers. Additionally, circulating biomarkers associated with myocardial fibrosis (including PIIINP, Galectin-3, and sST2) have emerged as promising indicators of cardiac remodeling and disease progression.

The STRIVE (Stratification Risk Via HF-QRS and Fibrosis Biomarkers in Heart Failure) Cohort is a prospective, multicenter observational study designed to systematically evaluate the prognostic significance of HF-QRS parameters and fibrosis biomarkers in patients with chronic heart failure (CHF).

Approximately 1500 patients with clinically stable CHF will be enrolled across multiple centers and followed for 18 months. Baseline data collection will include demographics, medical history, laboratory measures, standard echocardiographic parameters, HF-QRS signal analysis, and serum fibrosis biomarker levels (measured by ELISA). Clinical outcomes including cardiovascular death, first HF rehospitalization, malignant arrhythmia events, and all-cause rehospitalization will be prospectively recorded.

The study aims to assess the independent and incremental predictive value of HF-QRS and fibrosis biomarkers over traditional risk models. Furthermore, a multivariable prediction model integrating electrophysiological and molecular markers will be developed and internally validated to support dynamic risk stratification and personalized management strategies for CHF patients.

ELIGIBILITY:
Inclusion Criteria：

1. Age ≥18 years and ≤85 years
2. Diagnosis of chronic heart failure (CHF) based on ESC 2021 and AHA/ACC/HFSA 2022 guidelines
3. Presence of typical symptoms (e.g., exercise intolerance, dyspnea, orthopnea, paroxysmal nocturnal dyspnea, or fatigue) and signs (e.g., lower extremity edema, jugular venous distension, pulmonary rales)
4. Elevated NT-proBNP (>125 pg/mL, adjusted for BMI if >25 kg/m²)
5. Evidence of structural or functional cardiac abnormalities by echocardiography (LVEF ≤50%, E/e' >14, e' <9 cm/s, LV hypertrophy, or left atrial enlargement)
6. For HFpEF patients (LVEF ≥50%), at least one additional echocardiographic abnormality is required

The Main Exclusion Criteria:

1. End-stage renal disease requiring dialysis
2. Severe chronic pulmonary disease (e.g., moderate-to-severe COPD, pulmonary fibrosis)
3. Active malignancy or life expectancy <1 year
4. Severe anemia (Hb <8 g/dL) or uncontrolled thyroid dysfunction

4. Cardiogenic shock or need for mechanical ventilatory support 5. Severe cognitive impairment, psychiatric illness, or inability to comply with study procedures 6. Other non-cardiac causes that may mimic heart failure symptoms (e.g., advanced liver cirrhosis)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-85 years diagnosed with chronic heart failure (CHF), classified into HFrEF, HFmrEF, and HFpEF according to LVEF, receiving guideline-directed medical therapy (GDMT).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Cardiovascular mortality, First Heart Failure-related Rehospitalization, Malignant Arrhythmia, and All-Cause Rehospitalization | Up to 18 months
  A composite outcome including cardiovascular mortality, first heart failure-related rehospitalization, malignant arrhythmia events (ventricular tachycardia, ventricular fibrillation, torsades de pointes), and all-cause rehospitalization, assessed during the 18-month follow-up period.
All-Cause Mortality | Up to 18 months
  Death from any cause recorded during the 18-month follow-up period.

IPD SHARING:
Plan to Share IPD: No